CLINICAL TRIAL: NCT06330129
Title: Validity and Reliability of Trunk Muscle Strength Assessements With Isometric Dynamometry
Brief Title: Validity and Reliability of Trunk Strength Device
Acronym: PEGASUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: Balgrist Campus AG (Unknown)
Responsible Party: Principal Investigator, Jacopo Vitale, Principal Investigator, Schulthess Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pegasus01_Val
Record Dates: First submitted 2024-03-04; First posted 2024-03-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Trunk Muscle Strength
Keywords: Trunk muscle strength; Isometric device; Pegasus; Validity; Reliability; Muscle Activation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy subjects (Experimental): 30 healthy subjects undergo trunk muscle strength assessement using the Pegasus device, with repeated measurements to evaluate repeatability and correlation with both surface electromyography (EMG) and MRI scans of trunk muscles.
  Interventions: Device: CTT Pegasus

INTERVENTIONS:
Device: CTT Pegasus — The intervention aims to assess the construct validity of trunk flexor, extensor, and rotator muscle strength using the CTT PEGASUS isometric dynamometer (Leipzig, Germany). This involves correlating muscle strength measured isometrically with its physiological determinants: MRI-based anatomical cross-sectional area (CSA) in the lumbar region and muscle activation measured via surface electromyography (EMG) of spine and trunk muscles. Additionally, the intervention will assess the test-retest reliability of isometric strength of trunk flexors, extensors, and rotators.

SUMMARY:
The study aims to evaluate the accuracy and consistency of assessing trunk muscle strength using an isometric device (Pegasus, Leipzig, Germany). Thirty healthy volunteers will undergo maximal isometric strength testing with the device, repeated one week later to assess repeatability. Surface electrodes will measure muscle activation, while MRI scans will assess structural condition.

DETAILED DESCRIPTION:
The aim of the study is to assess the validity and repeatability of trunk muscle strength evaluation using an isometric device (Pegasus, Leipzig, Germany) and to investigate it. Thirty healthy volunteer participants will undergo testing of maximal isometric (non-moving) strength using this device. The same strength measurement procedure will be repeated one week later for all participants to determine if the measurements are repeatable, i.e., if the device is capable of providing similar strength data in two closely timed measurements. To assess whether the device actually provides reliable strength data for the trunk muscles, surface electrodes will be additionally placed on the involved muscles to understand the extent of neural activation of these muscles during the test. Additionally, an MRI examination will be conducted for all study participants to assess the structural condition of the trunk muscles.

ELIGIBILITY:
Inclusion Criteria:

* both male and female subjects
* age between 18 and 59 years
* BMI < 30 kg/m2
* cognitively intact (self-reported)
* autonomous walking

Exclusion Criteria:

* age under 18 years or over 60 years
* any prior spinal surgery or other musculoskeletal surgery having an impact on movement
* acute or chronic back pain in the last 6 months(self-reported)
* pregnancy (self-reported)
* inability to perform the planned set of activities included in the study (e.g. maximal voluntary contraction torque test)
* inability to give consent

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is open to both males and females (biologically); 15 for each group
Enrollment: 30 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
maximal isometric trunk muscle strength | 1 hour
  The computer-assisted test and trainig device (CTT) PEGASUS provides data on back muscle strength in isometric conditions, which constitutes the main endpoint of the present project.

SECONDARY OUTCOMES:
MRI muscle morphology | 0.5-1hour
  the anatomical crosssectional area (CSA) of trunk muscles (multifidus, erector spinae, rectus abdominis, and obliquus externus abdominis) evaluated through an abdominal MRI.
Electromyography (EMG) activity | 1hour
  the root mean square EMG activity recorded during maximal and submaximal voluntary contractions of respective muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland